CLINICAL TRIAL: NCT02868827
Title: Cholecalciferol Supplementation in Critically Ill Patients With Severe Vitamin D Deficiency in Intensive Care Unit- A Randomized Controlled Trial.
Brief Title: Cholecalciferol Supplementation in Critically Ill Patients With Severe Vitamin D Deficiency.
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The initial plan was 2 years but due to slow recruitment. We were able to screen 635 patients in 4 years and recruited only 127 patients.
Sponsor: King Abdullah Medical City (Other Government)
Responsible Party: Principal Investigator, Asiah Rugaan, Consultant and Head of Department - Intensive Care Unit, King Abdullah Medical City
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 16-252
Record Dates: First submitted 2016-08-07; First posted 2016-08-16 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Vitamin D Deficiency; Critical Illness
Keywords: cholecalciferol and critical illness; Mortality and cholecalciferol supplementation
MeSH Terms: conditions — Vitamin D Deficiency; Critical Illness | interventions — Cholecalciferol; Milk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cholecalciferol (Experimental): This group of patients will receive single high dose of vitamin D (Cholecalciferol) dissolved in 45 ml of fresh milk (Nestle)
  Interventions: Drug: Cholecalciferol
- Placebo (Placebo Comparator): This group of patients will receive placebo - 45 ml of fresh milk (Nestle) so that the amount, color, smell, taste etc will be the same as that of experimental drug)
  Interventions: Other: Milk (Nestle)

INTERVENTIONS:
Drug: Cholecalciferol — 400000 international Units of cholecalciferol will be dissolved in 45 ml of fresh milk (Nestle) and it will be given to interventional group patients through enteral route within 24 hours of ICU admission as a single dose.
  Other Names: Vitamin D3
  Arms: Cholecalciferol
Other: Milk (Nestle) — 45 ml of Nestle milk will given to patients assigned as placebo
  Arms: Placebo

SUMMARY:
The purpose of the research study is to determine whether a single high dose of vitamin D is helpful in reducing critical illness related complications in intensive care patients who are having sever vitamin D deficiency.

Vitamin D deficiency is quite common in critically ill patients ranging from 81.5% to 99%. A number of scientific studies have documented a strong correlation between low levels of vit.D and increased rate of adverse outcomes including infection, acute kidney injury and mortality in ICU patients. A recent randomized controlled trial (RCT) has demonstrated a 50% reduction in hospital mortality in severe vit.D deficient patients following a single high dose of cholecalciferol (Vitamin D3). However, the role of Vit.D supplementation to boost up host immune system and eventually reduction of mortality has yet to be determined by large randomized controlled trials in humans. Hence the study aims to run a randomized controlled trial (RCT) in order to study the role of Vitamin D in critically ill patients.

DETAILED DESCRIPTION:
DETAILED DESCRIPTION

Introduction: Vitamin D is a fat soluble vitamin and it affects multiple systems of our body. It not only plays a key role in musculoskeletal system but also works on our immune and cardiovascular systems. Because of its wide range of anti-inflammatory and metabolic properties, vitamin D, recently, has gained an immense importance among the intensivists.

Most of the critically ill patients have vitamin D deficiency and are at high risk of complications ranging from systemic inflammatory response syndrome (SIRS), sepsis, septic shock, multi-organ dysfunction, multi-organ failure and finally death. Immune system dysregulation has been thought to play a pivotal role in the development of sepsis. Onset and progression of sepsis are dependent upon a fine balance between pro-inflammatory and anti-inflammatory mediators of the immune system. Massive and uncontrolled release of pro-inflammatory cytokines leads to widespread tissue damage and multi-organ failure. It has been found that the cells of the immune system (both innate and acquired) express receptors for vitamin D. Low levels of it renders the immune system regulatory cells dysfunctional and in turn, increases the risk of infections and other adverse outcomes. It has been estimated that even with optimal treatment anywhere from 16% to more than 80% of patients with sepsis don't survive.

To improve the survival of critically ill patients, several research studies have been focused on the identification of various biomarkers and their correlation with disease severity. Timely supplementation of cholecalciferol has been demonstrated as one of the mortality reduction interventions. In recent studies, vitamin D has been identified as an important regulator of our immune system and its deficiency is quite common in ICU patients ranging from 81.5% to 99%.

A number of scientific studies have documented a strong correlation between low levels of vit.D and increased rate of adverse outcomes including infection with multi drug resistant organisms, acute kidney injury, decreased left ventricular ejection fraction and mortality in ICU patients. It has been found that the emergence of acinetobacter baumannii infections in significantly more common in vit D deficient critically ill patients and vit D deficiency is an independent risk factor for the development of Acinetobacter baumannii infections in intensive care unit.

A recent RCT has demonstrated 50% reduction in hospital mortality in patients with severe vit.D deficiency following a single high dose of cholecalciferol (Vitamin D3). However, the role of Vit.D supplementation to boost up host immune system and eventually reduction of mortality has yet to be determined by large randomized controlled trials.

In patients with severe vitamin D deficiency, gastrointestinal absorption of vit.D, after enteral supplementation could be variable depending upon the patient's gastrointestinal functions, critical illness and the activity of hepatic cytochrome P 450 system. In order to restore optimal vit.D level in critically ill patients (possibly within first 48 hours), a single high dose of it has been suggested on admission to ICU. As in critically ill patients, it is highly unlikely to restore Vitamin D within a reasonable period of time by supplementing 400-4000 international units/day (recommended daily allowance). Moreover, a single large dose of vit.D through the enteral route is highly unlikely to cause vit.D toxicity. The acutely toxic level of vit.D is considered to be more than 150 ng/ml. Furthermore, this high loading dose of cholecalciferol has been justified based on the safety findings of previous studies.

In addition, during a pilot study followed by a large randomized controlled trial conducted by Karen A et al, no serious adverse events were noted with a single high dose (540,000 I.U) of cholecalciferol. The highest 25-hydroxyvitamin D level measured was 107 ng/ml which is far below the currently suggested toxic level of vit.D (that is more than 150 ng/ml). Moreover, one patient in vitamin D3 group was found to have a total serum calcium level of 12 mg/dl and an ionized serum calcium level of 6 mg/dl but that patient had primary hyperparathyroidism (although normocalcemic at study inclusion). However, the incidence of falls and fracture was similar in vitamin D3 and placebo groups for a follow-up period of six months. So a single high dose of cholecalciferol is less likely to increase the incidence of hypocalcemia, hypercalciuria, falls and fractures which have been found to be increased with annual high doses of vitamin D3.

Hence the investigator intends to use a single high dose of cholecalciferol in order to restore it deficiency quickly, hopefully within 1 to 2 days in order to give maximum benefits to our critically ill patients right from the start of their illness.

The aim of our RCT is to study the role of Vit.D supplementation in critically ill patients. By boosting up the already struggling immune system of critically ill patients, the investigator assumes a significant reduction in mortality and other adverse outcomes.

Hypothesis: A single high dose of cholecalciferol supplementation improves survival in critically ill patients with severe vitamin D deficiency.

Null Hypothesis: A single high dose of Cholecalciferol supplementation in critically ill patients will not reduce the mortality and adverse outcomes.

Recruitment and randomization: Patients or their surrogates will be contacted on admission to ICU and study information will be provided to them by the research staff members. Consented patients will be randomized. Randomization list will be prepared by King Abdullah Medical City (KAMC) research center. The list will be used to prepare sealed envelopes each containing the assigned treatment. These envelopes will be stored in the pharmacy and opened up by the research pharmacist who will prepare medication/placebo for the randomized patients.

Blinding: Blinding will be done by research pharmacist in KAMC pharmacy. Fresh milk will be used as a placebo. The study medication (a white-colored, powdered form of cellulose based vit.D) will be dissolved in fresh milk so that both interventional drug and placebo will have the same color, odor, consistency, taste, and amount as that of interventional medication.

For all vit. D deficient patients, supplement 50,000 IU of cholecalciferol per week through the enteral route as a part of routine ICU treatment plan. As our recruited patients will be having severe vitamin D deficiency (Vit. D level below 12ng/ml) so both interventional and placebo group patients will receive our routine treatment for vit.D deficiency which is 50,000 IU of cholecalciferol through enteral route per week.

Intervention: Patients randomized to vitamin D group will receive 400,000 IU of cholecalciferol dissolved in 45 ml of fresh milk through orogastric tube/nasogastric tube/Oral within 1st 24 hours of ICU admission. This high dose is in addition to our routine treatment for vitamin D deficiency.

Post-recruitment retention strategies: the study will follow our patients for 30 days or as long as they stay in ICU after supplementation of a single high dose of vitamin D or placebo. As the investigators are working with critically ill patients, expecting at least a few weeks of hospital stay. However, the patient having early and quick recovery will be discharged home and will be followed up by one of the assigned research team members who will be contacting them by phone and inquire about any complications related to the research study.

Method: the investigator will complete a randomized controlled trial by supplementing cholecalciferol 400,000 IU versus placebo within 24 hours of ICU admission that would be added to our routine treatment for vit.D deficiency. Safety of this high dose of vit D has been validated in previous studies. This trial will employ block randomization and intention to treat protocol. This single-center study would be completed over a period of 2 complete years here in KAMC Intensive care Unit.

Laboratory Measurements: Blood samples will be obtained at baseline (day 0) and days 1, 3, 7, and 28 to assess serum parathyroid hormone, total and bioavailable 25-hydroxyvitamin D levels, phosphate, procalcitonin, leukocytic count, hemoglobin, creatinine, bilirubin, beta natriuretic peptide (BNP), blood glucose and albumin levels. In addition, the investigator will also measure urinary calcium and urinary creatinine levels

Data Collection: Patients will be followed up (1 month) closely for the development of study-drug related complications if any, for example, hypercalcemia, hypercalciuria, fractures, etc. Data elements to be collected will include, but not limited to:

1. - Date and time of admission to hospital
2. - Mode of admission (Emergency Room or in-patients)
3. - Date and time of ICU admission
4. - 25 - hydroxyl vitamin D level on admission to ICU.
5. - Sequential Organ Failure Assessment (SOFA) score
6. - Acute Physiology And Chronic Health Index (APACHI) Score 7-Patient's co-morbidities (Diabetes, Hypertension, Chronic kidney disease, Chronic obstructive pulmonary disease, Ischemic Heart Disease, Coronary Artery Bypass Grafting, Cerebrovascular accident, Arrhythmias, Anemias, smoking, obesity, cancer)

8 - Mode of Oxygen delivery to the patient 9 - Previous positive cultures and antibiotic therapy within the last 3 months 10 - Empirical antibiotic therapy on admission to hospital and ICU 11 - Baseline clinically relevant investigation, for example, Echo, Electrocardiography, Ultrasound Doppler for Deep venous thrombosis, CT brain/chest/abdomen, 12 - Endo/bronchoscopic findings if any 13 - Vasopressors and ionotropic support duration 14 - Central venous catheter, arterial line, pigtail, chest tube (site, date and time of insertion) 15 - Evidence of acute or acute on chronic kidney injury on admission to ICU. 16 - Surgeries - previous and recent surgeries and any post-op complications 17 - Previous immunosuppressive therapies for example chemo/radio/glucocorticoid therapy.

Sample size calculation: A recent RCT demonstrated almost 50% reduction in hospital mortality (46.1% in placebo versus 28.6% in Vit D group) by supplementing 540,000 IU of Vit D3 to critically ill patients having severe vitamin D deficiency (25-hydroxyvitamin D level ≤ 12 ng/ml). With an alpha = 5% (two tailed test), power = 95%, baseline mortality control group 30% and test group mortality 15%, the sample size required would be 195 patients per group. To account for losses to follow up of around 10%, the study aims to recruit 215 patients in each group. So the total number of patients required for both the groups would be 430 in 2 full years.

Statistical Analysis: the investigator will use an intention to treat approach to avoid the effects of crossover and dropout. Standard statistical analysis will include normally or near normally distributed variables reported as means and non-normally distributed variables as medians. Means will be compared by using student's t-test and medians by using Mann-Whitney U test. Differences in proportions among categorical data will be assessed using Fisher's exact test. A p-value of less than 0.05 will be considered to represent statistical significance for all comparisons.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older.
2. Both male and female
3. Within 24 hours from admission.
4. Having 25 -Hydroxyvitamin D level of 12 ng/ml or lower.

Exclusion Criteria

1. Pregnant or lactating females.
2. Do not resuscitate (DNR) status or comfort measures only
3. No consent
4. Severely impaired gastrointestinal functions (e.g, paralytic ileus, continuous nasogastric tube drainage, strict nil per oral- no medication, malabsorption syndrome, chronic diarrhea etc)
5. History of renal stones within past year
6. Past history of hypercalcemia, tuberculosis or sarcoidosis.
7. Baseline serum total calcium ≥10.6 mg/dl or ionized serum calcium ≥ 5.4 mg/dl.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2017-08-27 (Actual); Primary Completion 2019-11-09 (Actual); Study Completion 2019-11-09 (Actual)

PRIMARY OUTCOMES:
Reduction in hospital mortality | 28 days
  as assessed by hospital mortality rate

SECONDARY OUTCOMES:
Emergence of Multidrug resistant (MDR) organisms | 28 days
  as evidenced by microbiological culture and sensitivity reports from samples taken from patients blood, sputum,urine and body fluids.
Vasopressor requirement | 28 days
  as evidenced by invasive blood pressure monitoring during ICU stay.
Ventilator free days | 28 days
  How long is the free days
ICU length of stay | 28 days
  How long the patient will stay in ICU
Hospital length of stay | 28 days
  How long the patient will stay in Hospital
New onset of Acute kindney injury | 28 days
  It will be assessed by rising serum creatinine level and decreasing urine out put per hour.
Development of acute CVA | 28 days
  as evidenced by neurological deficit and CT sacn/MRI findings
Upper and lower GI bleeding | 28 days
  It will be assessed by decreasing hemoglobin levels and endoscopic findings.
Acute co-morbidities | 28 days
  including, acute kidney injury, Myocardial Infarction, Cerebrovascular accidents, upper or lower gastro intestinal bleed)

CONTACTS AND LOCATIONS:
Overall Officials: Asiah S Rugaan, MD, MRCP, Study Chair — King Abdullah Medical City Makkah
Locations (1):
- King Abdullah Medical City, Holy Capital, Mecca, Makkah Western, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Perron RM, Lee P. Efficacy of high-dose vitamin D supplementation in the critically ill patients. Inflamm Allergy Drug Targets. 2013 Aug;12(4):273-81. doi: 10.2174/18715281113129990047. PMID 23782210
- [Background] Quraishi SA, De Pascale G, Needleman JS, Nakazawa H, Kaneki M, Bajwa EK, Camargo CA Jr, Bhan I. Effect of Cholecalciferol Supplementation on Vitamin D Status and Cathelicidin Levels in Sepsis: A Randomized, Placebo-Controlled Trial. Crit Care Med. 2015 Sep;43(9):1928-37. doi: 10.1097/CCM.0000000000001148. PMID 26086941
- [Background] Higgins DM, Wischmeyer PE, Queensland KM, Sillau SH, Sufit AJ, Heyland DK. Relationship of vitamin D deficiency to clinical outcomes in critically ill patients. JPEN J Parenter Enteral Nutr. 2012 Nov;36(6):713-20. doi: 10.1177/0148607112444449. Epub 2012 Apr 20. PMID 22523178
- [Background] Lee P, Eisman JA, Center JR. Vitamin D deficiency in critically ill patients. N Engl J Med. 2009 Apr 30;360(18):1912-4. doi: 10.1056/NEJMc0809996. No abstract available. PMID 19403914
- [Background] Matthews LR, Ahmed Y, Wilson KL, Griggs DD, Danner OK. Worsening severity of vitamin D deficiency is associated with increased length of stay, surgical intensive care unit cost, and mortality rate in surgical intensive care unit patients. Am J Surg. 2012 Jul;204(1):37-43. doi: 10.1016/j.amjsurg.2011.07.021. Epub 2012 Feb 10. PMID 22325335
- [Background] Braun A, Chang D, Mahadevappa K, Gibbons FK, Liu Y, Giovannucci E, Christopher KB. Association of low serum 25-hydroxyvitamin D levels and mortality in the critically ill. Crit Care Med. 2011 Apr;39(4):671-7. doi: 10.1097/CCM.0b013e318206ccdf. PMID 21242800
- [Background] Braun AB, Litonjua AA, Moromizato T, Gibbons FK, Giovannucci E, Christopher KB. Association of low serum 25-hydroxyvitamin D levels and acute kidney injury in the critically ill. Crit Care Med. 2012 Dec;40(12):3170-9. doi: 10.1097/CCM.0b013e318260c928. PMID 22975885
- [Background] Arnson Y, Gringauz I, Itzhaky D, Amital H. Vitamin D deficiency is associated with poor outcomes and increased mortality in severely ill patients. QJM. 2012 Jul;105(7):633-9. doi: 10.1093/qjmed/hcs014. Epub 2012 Feb 12. PMID 22331959
- [Background] Braun AB, Gibbons FK, Litonjua AA, Giovannucci E, Christopher KB. Low serum 25-hydroxyvitamin D at critical care initiation is associated with increased mortality. Crit Care Med. 2012 Jan;40(1):63-72. doi: 10.1097/CCM.0b013e31822d74f3. PMID 21926604
- [Background] Turkoglu M, Aygencel G, Dizbay M, Tuncel AF, Arslan Candir B, Deligoz Bildaci Y, Pasaoglu H. Is vitamin D deficiency associated with development of Acinetobacter baumannii infections in critically ill patients? J Crit Care. 2013 Oct;28(5):735-40. doi: 10.1016/j.jcrc.2013.03.017. PMID 24018297
- [Background] Amrein K, Schnedl C, Holl A, Riedl R, Christopher KB, Pachler C, Urbanic Purkart T, Waltensdorfer A, Munch A, Warnkross H, Stojakovic T, Bisping E, Toller W, Smolle KH, Berghold A, Pieber TR, Dobnig H. Effect of high-dose vitamin D3 on hospital length of stay in critically ill patients with vitamin D deficiency: the VITdAL-ICU randomized clinical trial. JAMA. 2014 Oct 15;312(15):1520-30. doi: 10.1001/jama.2014.13204. PMID 25268295
- [Background] Spriet I, Meersseman W, de Hoon J, von Winckelmann S, Wilmer A, Willems L. Mini-series: II. clinical aspects. clinically relevant CYP450-mediated drug interactions in the ICU. Intensive Care Med. 2009 Apr;35(4):603-12. doi: 10.1007/s00134-008-1383-2. Epub 2009 Jan 9. PMID 19132344
- [Background] Michaud J, Naud J, Ouimet D, Demers C, Petit JL, Leblond FA, Bonnardeaux A, Gascon-Barre M, Pichette V. Reduced hepatic synthesis of calcidiol in uremia. J Am Soc Nephrol. 2010 Sep;21(9):1488-97. doi: 10.1681/ASN.2009080815. Epub 2010 Jul 1. PMID 20595682
- [Background] McNally JD. Vitamin D as a modifiable risk factor in critical illness: questions and answers provided by observational studies. J Pediatr (Rio J). 2014 Mar-Apr;90(2):99-101. doi: 10.1016/j.jped.2013.12.002. Epub 2013 Dec 19. No abstract available. PMID 24361295
- [Background] Amrein K, Sourij H, Wagner G, Holl A, Pieber TR, Smolle KH, Stojakovic T, Schnedl C, Dobnig H. Short-term effects of high-dose oral vitamin D3 in critically ill vitamin D deficient patients: a randomized, double-blind, placebo-controlled pilot study. Crit Care. 2011;15(2):R104. doi: 10.1186/cc10120. Epub 2011 Mar 28. PMID 21443793
- [Background] Bacon CJ, Gamble GD, Horne AM, Scott MA, Reid IR. High-dose oral vitamin D3 supplementation in the elderly. Osteoporos Int. 2009 Aug;20(8):1407-15. doi: 10.1007/s00198-008-0814-9. Epub 2008 Dec 20. PMID 19101755
- [Background] von Restorff C, Bischoff-Ferrari HA, Theiler R. High-dose oral vitamin D3 supplementation in rheumatology patients with severe vitamin D3 deficiency. Bone. 2009 Oct;45(4):747-9. doi: 10.1016/j.bone.2009.06.012. Epub 2009 Jun 17. PMID 19539796
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Background] Vieth R. Critique of the considerations for establishing the tolerable upper intake level for vitamin D: critical need for revision upwards. J Nutr. 2006 Apr;136(4):1117-22. doi: 10.1093/jn/136.4.1117. PMID 16549491
- [Background] Sanders KM, Stuart AL, Williamson EJ, Simpson JA, Kotowicz MA, Young D, Nicholson GC. Annual high-dose oral vitamin D and falls and fractures in older women: a randomized controlled trial. JAMA. 2010 May 12;303(18):1815-22. doi: 10.1001/jama.2010.594. PMID 20460620
- [Background] Smith H, Anderson F, Raphael H, Maslin P, Crozier S, Cooper C. Effect of annual intramuscular vitamin D on fracture risk in elderly men and women--a population-based, randomized, double-blind, placebo-controlled trial. Rheumatology (Oxford). 2007 Dec;46(12):1852-7. doi: 10.1093/rheumatology/kem240. Epub 2007 Nov 12. PMID 17998225